CLINICAL TRIAL: NCT03931668
Title: A Single Site, Randomized, Double-blind, Placebo-controlled, Incremental Phase I Clinical Trial: to Evaluate the Tolerance, PK and PD Effects of TPN-672 Maleate in Chinese Healthy Volunteers After Single Dose Administration.
Brief Title: Tolerance, PK and PD Effects Study of TPN-672 in Chinese Healthy Volunteers
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Jiangsu Kanion Pharmaceutical Co. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: SMHC-180; TPN672-KYHY-201801 (Other: Kanion Pharmaceutical)
Record Dates: First submitted 2019-04-13; First posted 2019-04-30 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-04

CONDITIONS: PHA1A
Keywords: tolerance; pharmacokinetics; pharmacodynamics; TPN-672

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 0.125mg single dose (Experimental): single dose of TPN-672 0.125mg, 2 subjects
  Interventions: Drug: TPN-672
- 0.25mg single dose (Experimental): single dose of 0.25mg, 10 subjects (8 for TPN-672, 2 for placebo)
  Interventions: Drug: TPN-672
- 0.5mg single dose (Experimental): single dose of 0.5mg, 10 subjects (8 for TPN-672, 2 for placebo)
  Interventions: Drug: TPN-672
- 1mg single dose (Experimental): single dose of 1mg, 10 subjects (8 for TPN-672, 2 for placebo)
  Interventions: Drug: TPN-672
- 2mg single dose (Experimental): single dose of 2mg, 10 subjects (8 for TPN-672, 2 for placebo)
  Interventions: Drug: TPN-672
- 3mg single dose (Experimental): single dose of 3mg, 10 subjects (8 for TPN-672, 2 for placebo)
  Interventions: Drug: TPN-672
- 4mg single dose (Experimental): single dose of 4mg, 10 subjects (8 for TPN-672, 2 for placebo)
  Interventions: Drug: TPN-672

INTERVENTIONS:
Drug: TPN-672 — single dose of TPN-672 maleate tablet
  Other Names: TPN-672 maleate tablet

SUMMARY:
This is a single-site, randomized, double-blind, placebo-controlled, incremental phase I clinical trial to evaluate preliminarily the tolerance, pharmacokinetics and pharmacodynamic effects of TPN672 maleate in Chinese healthy volunteers after single dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Body weight > 50kg(male) or > 45kg(female), 19 <BMI<26 kg/m2.
* Good communication with investigators, willingness and ability to abide by the lifestyle restrictions stipulated in clinical trial
* Women or men within childbearing age do not have a fertility plan within 3 months after the end of the trial, and agree to adopt contraceptive measures approved (such as intrauterine device, condom, sperm killing gel, condom, uterine cap, etc.) throughout the clinical trial period.
* Fully understand the purpose and requirements of the trial, voluntarily participate in the clinical trial and sign the written informed consent, can complete the entire trial process according to the requirements of the trial.

Exclusion Criteria:

* Investigator determined that there were diseases or functional disorders affecting clinical trials, including, but not limited to, central nervous system, cardiovascular system, respiratory system, digestive system, urinary system, endocrine system and blood system.
* Mental illness or previous history of mental illness;
* Have a history of ophthalmic diseases, such as abnormal color vision, retinitis pigmentosa, macular degeneration, etc.
* Have a history of malignant tumors or other diseases that are not suitable for clinical trials;
* Any surgical condition or condition that may significantly affect drug absorption, distribution, metabolism and excretion, or that may pose a hazard to the subjects participating in the study, such as history of gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), urinary tract obstruction or dysuria, gastroenteritis, gastrointestinal ulcer, gastrointestinal bleeding, etc.
* Those who are known to have a history of drug allergy, allergic disease or allergic constitution of the tested drug ingredients or similar drugs;
* Smokers who smoked more than 10 cigarettes or the same amount of tobacco per day in the first year of screening;
* Alcohol addiction within 1 year before screening, with an average weekly alcohol intake of more than 14 units (1 unit = 285 ml beer or 25 ml spirits or 150 ml wine) or positive alcohol breath test;
* Those who had a history of drug abuse or drug abuse within 1 year before screening, or those who had positive urinary drug screening;
* Physical examination, current medical history and vital signs were found to be abnormal by researchers and have clinical significance.
* Resting pulse rate < 55/min or > 100/min; systolic pressure < 90 mmHg or > 140 mmHg, diastolic pressure < 60 mmHg or > 90 mmHg;
* 12-lead electrocardiogram (ECG) examination was found to be abnormal by investigator and had clinical significance; or the following ECG abnormalities occurred: PR interval > 220 ms, QRS complex wave duration > 120 ms, long QT syndrome (QTc > 450 ms);
* Family history of sudden cardiac death (less than 40 years old);
* Abnormal blood routine examination and urine routine examination have clinical significance.
* Aspartate transferase (AST), alanine transferase (ALT), creatinine (Cr), urea nitrogen (BUN) exceeded the normal upper limit.
* HBsAg, HCV-Ab, HIV-Ab and TRUST positive patients;
* Pregnant or lactating women or male subjects whose spouses have child-rearing plans within three months;
* Those who took any medicine within 2 weeks before admission, including prescription and non-prescription drugs;
* Blood donation or blood loss (> 200 ml) within 3 months before admission, or a history of using blood products;
* Participated in any clinical trials within 3 months before admission;
* Those who had a history of operation within 3 months before admission, or who had not recovered from the operation, or who had anticipated operation plan during the trial period;
* Do not agree to abide by the following conditions during the experiment: prohibit the use of tobacco, alcohol or caffeine-containing beverages, avoid strenuous exercise;
* Personnel directly related to this clinical trial;
* Investigator believes that other subjects are not suitable for the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 62 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-10-17 (Estimated); Study Completion 2020-12-17 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 48 hours
  Number of Subjects with adverse events during clinical trial
Cmax | 48 hours
  Maximum Plasma Concentration
AUC | 48 hours
  Area Under the Curve
Tmax | 48 hours
  Time to Cmax
T1/2 | 48 hours
  Time of half life
ACR | 48 hours
  Apparent Clearance Rate
ADV | 48 hours
  Apparent Distribution Volume

SECONDARY OUTCOMES:
prolactin | 48 hours
  serum prolactin test
temperature | 48 hours
  ear temperature
pulse rate | 48 hours
  pulse rate
respiratory | 48 hours
  frequency of respiratory per minute
blood pressure | 48 hours
  lying blood pressure， systolic and diastolic
electrocardiogram(ECG) | 48 hours
  the number of subjects with abnormal ECG report by 12-lead electrocardiogram
QTc | 48 hours
  QTc interval
Extrapyramidal symptoms | 48 hours
  Simpson Angus Rating Scale (SAS), total score ranges from 0 to 40, of which lower values represent a better outcome.
Involuntary Movement | 48 hours
  Abnormal Involuntary Movement Scale (AIMS), total score ranges from 0 to 14, of which lower values represent a better outcome.
Akathisia | 48 hours
  Barnes Akathisia Rating Scale (BARS), total score ranges from 0 to 40, of which lower values represent a better outcome.
IL-6 | 48 hours
  Serum concentration of Interleukin-6
IL-4 | 48 hours
  Serum concentration of Interleukin-4
IL-1 | 48 hours
  Serum concentration of Interleukin-1
IL-2 | 48 hours
  Serum concentration of Interleukin-2
INF-gamma | 48 hours
  Serum concentration of Interferon-gamma
TNF-alpha | 48 hours
  Serum concentration of Tumor necrosis factor-alpha
5-HT | 48 hours
  Serum concentration of serotonin
DA | 48 hours
  Serum concentration of Dopamine
NE | 48 hours
  Serum concentration of Norepinephrine
BDNF | 48 hours
  Serum concentration of Brain-derived neurotrophic factor
Glutamic acid | 48 hours
  Serum concentration of Glutamic acid
GABA | 48 hours
  Serum concentration of gamma-aminobutyric acid

CONTACTS AND LOCATIONS:
Overall Officials: Yifeng SHEN, MD PhD, Study Director — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No